CLINICAL TRIAL: NCT03769038
Title: Long-term Outcomes of Successful Chronic Total Occlusion Percutaneous Coronary Interventions Using the Antegrade and Retrograde Dissection and Re-entry Approach
Brief Title: Antegrade and Retrograde Dissection and Re-entry Approach for CTO
Acronym: LOTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJYY-LL-FJ-059
Record Dates: First submitted 2018-11-07; First posted 2018-12-07 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2021-10

CONDITIONS: Chronic Total Occlusion of Coronary Artery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic Total Occlusion and Restenosis (Other): contemporary antegrade or retrograde dissection and re-entry (ADR or RDR) to open CTO
  Interventions: Device: chronic total occlusion

INTERVENTIONS:
Device: chronic total occlusion — chronic total occlusion of coronary atery was opened and then stents were placed

SUMMARY:
BACKGROUND：Chronic total occlusion (CTO) angioplasty is one of the most challenging procedures remaining for the interventional operator. Today, with contemporary CTO negotiation available strategies and significant operator expertise, the literature reports a 50%-95% success rate for recanalizing CTOs. But PCIs of CTO lesions still carry a high rate of in-stent restenosis (ISR). Because previous reports have not specifically compare contemporary antegrade and retrograde dissection and re-entry dissection (ADR/RDR) technique on the long-term impact of ISR, so the investigators focused on the objective.

OBJECTIVES: This study hope to evaluate the frequency of angiographic ISR and further elucidate some ISR related higher risk factors among CTO PCI patients in intimal stent group using antegrade or retrograde wire escalation (AWE/RWE) techniques and sub-intimal stent group using contemporary antegrade or retrograde dissection and re-entry (ADR and/or RDR).

METHODS: A total of 300 consecutive selected patients with CTO lesion who will undergo successful revascularization by AWE/RWE and ADR/RDR techniques treatment will be enrolled in this prospective multicenter registry from December 1 2018 to December 31 2019. The primary study endpoint of the protocol is the bionary in-stent restenosis of CTO vessels at angiographic follow-up about 13 months. The secondary endpoints are: 1) CTO technique and procedure success rate; and 2) in-hospital and 30 days MACE (Cardiac death, acute myocardial infarction, urgent repeat tratget vessel revascularization with either pericardiocentssis or surgery and stroke and stent thrombosis and stroke); 6months and 1-year and 2-year MACE including death, MI, and target CTO vessel revascularization and stroke ; and 3) Restenosis scores (R-scores) of related risk factors.

DETAILED DESCRIPTION:
METHODS

1. Trial overview and study population.

   ① This clinical trial is a prospective, exploratory, nonrandomized, multicenter trial evaluating the frequency of angiographic restenosis and clinical outcomes among patients undergoing CTO PCI in intimal stent group using antegrade or retrograde wire escalation (AWE/RWE) techniques and sub-intimal stent group using contemporary antegrade or retrograde dissection and re-entry (ADR or RDR) with everolimus-eluting stents (XIENCE Coronary Stent).

   ②According to high patient's volume registry studies in CTO lesions, the patients percentage of ADR or RDR strategy application was just only 20-25%36-37. If to get 60 patients for ADR or RDR strategies, the minimum CTO number are 300 patients. So in this registry study, 300 CTO cases, to which PCI will be attempted, are prospectively enrolled from Dec 1st 2018 to Dec 31st 2019 in the CTO registries of ten centers. The study was approved by the institutional review board at each site. For patients with multiple treated CTO, only the first CTO attempted was considered for the analysis.

   ③ Exclusions included age <18-years-old or >85-years-old, left ventricular ejection fraction ≦30%, allergy to medications (antiplatelet drugs, heparin, metal alloys, or contrast agents), a planned surgery within 6 months of PCI or planned thrombolysis, pregnant, a life expectancy of <6 months.

   ④ Participants will sign written informed consent for long-term telephone FU before the interventional procedure. Participants will be followed by a clinical visit or by a telephone interview for 30 day, 6 months and 12 months and 24 months post-procedure for assessment of adverse events. All patients with successful CTO PCI and without moderate or severe renal insufficiency will be scheduled for angiographic follow-up at 13 months. Compared with CTA, coronary angiography to evaluate restenosis is appropriate in all patients especially for severe coronary heart diseases patients with atrial fibrillation and ventricular arrhythmia. It could provide accurate information about mild-severe angulation lesion and the stents traits like total stent length. Procedural and outcome data collection will be collected and entered by operators entered into a dedicated database.

   ⑤ The study will be performed in accordance with the Declaration of FMMU.
2. Study endpoints and definitions The primary study endpoint of the protocol is the bionary in-stent restenosisof CTO vessels at the scheduled angiographic follow-up at 13 months. The secondary endpoints are: 1) CTO technique and procedure success rate; and 2) in-hospital and 30 days MACE (Cardiac death, acute myocardial infarction, urgent repeat tratget vessel revascularization with either pericardiocentssis or surgery and stroke and stent thrombosis and stroke); 6 months and 1-year and 2-year MACE including death, MI, and target CTO vessel revascularization and stroke ; and 3) Restenosis scores (R-scores) of related risk factors.

Coronary CTOs will be defined as angiographic evidence of total occlusions with TIMI (Thrombolysis In Myocardial Infarction) flow grade 0 and estimated durations of at least 3 months. Estimation of the occlusion duration is based on first onset of anginal symptoms, prior history of myocardial infarction in the target vessel territory, or comparison with a prior angiogram.

Procedural success will be defined as angiographic success(final residual stenosis <30% by visual estimation and TIMI flow grade 3 after CTO recanalization).

Clinical success will be defined as a procedural success without In-hospital MACCEs. In-hospital MACCEs is defined as the composite of non-Q-wave and Q-wave myocardial infarction (MI), recurrent angina requiring urgent repeat revascularization with PCI orcoronary bypass surgery, stroke, and death. Non-Q-wave MI is defined as creatine kinase-MB enzyme elevation >3 times the upper limit of normal. When new pathological Q waves, in addition to enzyme elevation, will be observed on the electrocardiogram, the event is defined as a Q-wave MI. In all patients, creatine kinase and creatine kinase-MB is evaluated 6 h after the procedure and until their normalization if levels is abnormal.

Lesion complexity will be judged using the J-CTO (20)and calculated by allocating 1 point each for non-tapered proximal cap (ie, blunt or ambiguous), any calcification, any tortuosity, occlusion length >20 mm and any prior unsuccessful attempt. J-CTO score of ≥2 was defined as complex.

CTO proximal cap location is defined according to American Heart Association (AHA) classification and additionally coded as either ostial or non-ostial and proximal (left main, proximal left anterior descending, proximal circumflex or proximal right coronary artery) or distal (all other sites). Cap morphology is coded as blunt or tapered, or as ambiguous when there is lack of clarity over the origin of the ongoing vessel. Calcification within the CTO is coded as none visible, mild(spots only), moderate (<50% of vessel circumference) or severe (>50% of vessel circumference). Disease proximal and distal to the CTO is classified as absent, mild, moderate or severe. Aproximal or distal cap side branch is considered present if occurring ≤3 mm from the respective CTO cap. Occlusion length is estimated by dual injection, or from apparent length after guidewire crossing. Collaterals are classified according to Cohen and Rentrop and deemed interventional if, on angiographic inspection, are thought amenable to crossing by a guidewire and a microcatheter by the operator.

All deaths are considered cardiac unless otherwise documented. Stent thrombosis is defined according to the Academic Research Consortium criteria (13). Reocclusionis defined as a TIMI flow grade of 0 to1in the target CTO vessel, where restenosis is defined as > 50% luminal narrowing at the segment site, including the stent and 5 mm proximal and distal to the stent edges. Target lesion revascularization (TLR) is defined as any repeat PCI or coronary artery bypass graft surgery of the target lesion that includes 5 mm proximal and distal to the stented vessel segment.

A procedure is considered retrograde if an attempt is made to cross the lesion through a collateral vessel supplying the target vessel distal to the lesion. Complex lesions with unclear location of the proximal cap or with poor distal target are initially attempted by the retrograde approach. In those cases, after positioning of a microcatheter at the distal CTO cap, a true-to-true retrograde lumen crossing technique is first attempted for shorter lesions (<20 mm). When entering in the subintimal space or with longer lesions, knuckled wires are used to reach the proximal cap, followed most often by reverse-controlled anterograde and retrograde re-entry techniques.

A procedure is considered antegrade if no retrograde crossing attempts are made. An anterograde approach is initially attempted for short lesions (<20 mm) with clear proximal cap location and good distal vessel target using a wiring strategy. Anterograde dissection/re-entry using dedicated devices (CrossBoss and Stingray catheters) is, however, preferred for longer lesions with an optimal distal re-entry zone, without significant side branches that could be occluded by the technique, or when an initial wire escalation strategy failed. Wire-based anterograde dissection/re-entry was also used successfully when an initial attempt at crossing from a "true-to-true" approach failed. Such a strategy involves the use of a microcatheter delivered on a knuckled polymer-jacketed wire advanced into the subintimal dissection plane, with subsequent re-entry into the true distal lumen using a stiff tapered guidewire or a knuckled guidewire. A Stingray system will be used to cross from the false lumen to the true lumen, the so-called hybrid procedure, rapidly switching from one approach to another when the initial strategy attempted is failing.

ELIGIBILITY:
Inclusion Criteria:

* CTO time >3months and CTO length >20mm

Exclusion Criteria:

* age <18-years-old or >85-years-old,
* left ventricular ejection fraction ≦30%,
* allergy to medications (antiplatelet drugs, heparin, metal alloys, or contrast agents),
* a planned surgery within 6 months of PCI or planned thrombolysis,

  * pregnant,
  * a life expectancy of <6 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
the bionary in-stent restenosis of CTO vessels at the scheduled angiographic follow-up at 13 months. | 13months after PCI
  the diamater of stents less than 50%

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of fourth military medical university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT03769038/Prot_SAP_000.pdf